CLINICAL TRIAL: NCT03345862
Title: Effectiveness of a Multi-component Non-pharmacological Intervention to Reduce the Social Isolation and Loneliness of Elderly Residents at Home
Brief Title: Effectiveness of a Intervention to Reduce the Social Isolation and Loneliness of Elderly Residents at Home
Acronym: ASyS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Luis Angel Perula de Torres, Dr. Ph., Andaluz Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AP-0079-2016
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Social Isolation, Loneliness (Descriptors Included in the MeSH)
Keywords: Social isolation, Loneliness, Health Related Quality of Life
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Non-pharmacological multicomponent intervention
  Interventions: Behavioral: non-pharmacological multicomponent
- Control (No Intervention): Not intervention, usual attention

INTERVENTIONS:
Behavioral: non-pharmacological multicomponent — Following the proposal of Nicholson & Shellman, (2013) collected in its CARELINK program, an intervention is proposed that includes: 6 sessions at home [30-60 minutes] for 16 weeks (1 fortnightly session) and 5 telephone sessions [20 min.] That will be intercalated (in the 16 weeks) depending on the particular characteristics of each person. The first visit, aimed at defining objectives and creating a relationship of trust for future visits.
  Arms: Intervention

SUMMARY:
* Objectives: To evaluate the effectiveness, in terms of reducing social isolation and improving the Health Related Quality of Life (HRQOL), of a non-pharmacological multicomponent intervention in elderly telecare users.
* Design: Clinical trial randomized by cluster, multicentric.
* Location: 14 health centers of the Andalusian Health Service (Spain).
* Subjects and methods: Subjects with social isolation. Age 65 or older. Residents in your home. Persons with cognitive impairment or dementia, difficulty in responding to scales, legal incapacitation or not giving consent will be excluded.

  9 health centers will be randomly assigned to the intervention and control groups. The people of both groups will be evaluated at baseline, at 4 and at 6 months. 57 subjects will be included in each group (n = 114).

Variables: a) Independent: of the professional and of the patients (sociodemographic, healthcare, morbidity, intervention performed -multicomponent vs. non-intervention-) b) Dependents: social support, loneliness and HRQoL.

The intervention includes 8 sessions at home [1 hour], every 15 days and 4 telephone [30 minutes] -1 monthly-. To measure the effectiveness of the intervention, the Duke-UNC Functional Social Support Questionnaire (DUFSS), the De Jong-Gierveld Scale of loneliness, and the EuroQol-5D will be used to measure HRQoL.

Univariate, bivariate and multivariate statistical analysis (multiple linear regression).

-Aspects ethico-legal: Standards of good clinical practice and ethical principles of the Declaration of Helsinki. Informed consent. Application for authorization to the management of the Sanitary District.

DETAILED DESCRIPTION:
-Subjects and methods: Subjects with social isolation. Age 65 or older. Residents in your home. Telecare users. Persons with cognitive impairment or dementia, difficulty in responding to scales, legal incapacitation or not giving consent will be excluded.

9 health centers will be randomly assigned to the intervention and control groups. The people of both groups will be evaluated at baseline, at 4 and at 6 months. 57 subjects will be included in each group (n = 114).

Variables: a) Independent: of the professional and of the patients (sociodemographic, healthcare, morbidity, intervention performed -multicomponent vs. non-intervention-) b) Dependents: social support, loneliness and HRQoL.

The intervention includes 6 sessions at home [30-60 minutes], every 15 days and 5 telephone [20 minutes] -1 monthly-. To measure the effectiveness of the intervention, the Duke-UNC Functional Social Support Questionnaire (DUFSS), the De Jong-Gierveld Scale of loneliness, and the EuroQol-5D will be used to measure HRQoL. Analysis by intention to treat. Univariate, bivariate and multivariate statistical analysis (multiple linear regression).

-Aspects ethico-legal: Standards of good clinical practice and ethical principles of the Declaration of Helsinki. Informed consent. Application for authorization to the management of the Sanitary District. Approval of the Ethics and Clinical Research Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older.
2. Residents in your home (not institutionalized).
3. Present social isolation: score less than 32 (social support perceived low) with the Duke-UNC Functional Social Support Questionnaire (DUFSS).

Exclusion Criteria:

1. Cognitive impairment (Mini-mental <22), or medical diagnosis of dementia.
2. Difficulty responding to measurement scales due to language barriers.
3. Legal incapacitation.
4. Do not grant consent for participation in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Social isolation | 6 months
  Duke-UNC Functional Social Support Questionnaire (DUFSS), which reflects the opinion on the availability of other people to offer help in difficulties, skills in social relations and empathic and emotional communication.
loneliness | 6 months
  De Jong-Gierveld de Soledad Scale, which assesses individual subjective perception of social participation or isolation in the elderly population.

SECONDARY OUTCOMES:
Health Related Quality of Life | 6 months
  Health Related Quality of Life (EuroQol-5D scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Angel Perula de Torres, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No